CLINICAL TRIAL: NCT00465946
Title: Effect of Dietary Salt Supplemantation in Vasovagal Syncope Prophylaxis: A Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HCPA04-071; HCPA04-071
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Healthy
Keywords: Salt supplementation; Vasovagal syncope; Orthostatic tolerance; Healthy volunteers
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Salt Supplementation

SUMMARY:
Syncope is a syndrome consisting of a relatively short period of temporary and self-limited loss of consciousness caused by transient diminution of blood flow to the brain (most often the result of systemic hypotension). The objective of this study was to evaluate the effect of salt supplementation in vasovagal syncope prophylaxis.

DETAILED DESCRIPTION:
Healthy volunteers without use of medicines with except contraceptives orals that met the exclusion criteria were consecutively enrolled in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Use medicines
* Previous diseases
* Incapacity of to understand and to sign the term consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-06; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the salt supplementation in the prophylaxis of the vasovagal syncope

SECONDARY OUTCOMES:
Evaluate the supplementation salt increases the orthostatic tolerance
Analyze the supplementation salt increases the plasmatic volume

CONTACTS AND LOCATIONS:
Overall Officials: Leandro I Zimerman, MD, Principal Investigator — Associate Professor
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: The Hospital of Clinics of Porto Alegre is a Public Company of Right Private member of the net of academical hospitals of Ministry of Education and linked academically to the Federal University of Rio Grande do Sul. — http://www.hcpa.ufrgs.br